CLINICAL TRIAL: NCT02373280
Title: A Prospective, Single-center, Open-label, Clinical Trial to Compare the 10-day Sequential Therapy and 7-day Culture Based Tailored Therapy for the Eradication of Helicobacter Pylori
Brief Title: The Efficacy of the 7 Days Tailored Therapy as the 1st Eradication of H. Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1407/259-005
Record Dates: First submitted 2015-02-05; First posted 2015-02-27 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Helicobacter Infection
Keywords: Helicobacter pylori; tailored therapy; eradication
MeSH Terms: conditions — Helicobacter Infections | interventions — Esomeprazole; Amoxicillin; Clarithromycin; Metronidazole; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Patients selected study
Oversight: Data Monitoring Committee: No

ARMS (4):
- 10 day sequential group (Active Comparator): After proving H. pylori infection, the participant will receive the empirical 10 day sequential regimen (Esomeprazole, nexium® 40 mg bid 10 days (D1-D10)+amoxicillin® 1 g bid 5 days (D1-D5)+clarithromycin, klaricid® 500mg bid 5 days (D6-D10)+metronidazole, flasinyl® 500mg tid 5 days (D6-D10) for treatment of H. pylori infection in this group.
  Interventions: Drug: 10 day sequential therapy (Esomeprazole, amoxicillin, clarithromycin, metronidazole)
- 7 days tailored PPI triple therapy group (Experimental): After proving H. pylori infection, the participant received endoscopic guided biopsy for H. pylori culture and MIC. Based on antimicrobial susceptibility testing, the participant will receive 7 day tailored regimen [PPI triple therapy (Esomeprazole, nexium® 40 mg bid 7 days (D1-D7)+amoxicillin® 1 g bid 7 days (D1-D7)+clarithromycin, klaricid® 500mg bid 7 days (D1-D7)] in this group.
  Interventions: Drug: 7 day tailored PPI triple therapy (clarithromycin-containing triple therapy)
- 7 days tailored MEA therapy group (Experimental): After proving H. pylori infection, the participant received endoscopic guided biopsy for H. pylori culture and MIC. Based on antimicrobial susceptibility testing, the participant will receive 7 day moxifloxacin triple therapy [Esomeprazole, nexium® 40 mg bid 7 days (D1-D7)+Moxifloxacin, avelox® 400 mg qd 7 days (D1-D7)+Amoxicillin® 1 g bid 7 days (D1-D7)] in this group.
  Interventions: Drug: 7 day moxifloxacin based triple therapy [Esomeprazole, Moxifloxacin, Amoxicillin]
- 7 or 14 days tailored EBMT therapy group (Experimental): After proving H. pylori infection, the participant received endoscopic guided biopsy for H. pylori culture and MIC. Based on antimicrobial susceptibility testing, the participant will receive 7 day bismuth quadruple therapy [Esomeprazole, nexium® 40 mg bid 7 days (D1-D7)+Tri potassium dicitrate bismuthate, denol® 300 mg qid 7 days (D1-D7)+Metronidazole, flasinyl® 500 mg tid 7 days (D1-D7)+Tetracycline® 500 mg qid 7 days (D1-D7)] in this group. If there was no metronidazole resistance, the treatment was 7 days in duration. If metronidazole resistance was evident, treatment duration was 14 days.
  Interventions: Drug: 7 or 14 days tailored EBMT therapy group (bismuth quadruple therapy)

INTERVENTIONS:
Drug: 10 day sequential therapy (Esomeprazole, amoxicillin, clarithromycin, metronidazole) — In this group, patients will receive the 10 day sequential regimen for eradication of H. pylori. 10 day sequential regimen is like follows; Esomeprazole 40 mg bid 10 days (D1-D10)+amoxicillin 1 g bid 5 days (D1-D5)+clarithromycin 500 mg bid 5 days (D6-D10)+metronidazole 500 mg tid 5 days (D6-D10).
  Arms: 10 day sequential group
Drug: 7 day tailored PPI triple therapy (clarithromycin-containing triple therapy) — the participants received PPI based triple therapy[Esomeprazole 40 mg bid 7 days (D1-D7)+amoxicillin 1000mg bid 7 days (D1-D7)+clarithromycin 500mg bid 7 days (D1-D7)]
  Other Names: 7d PPI triple therapy
  Arms: 7 days tailored PPI triple therapy group
Drug: 7 day moxifloxacin based triple therapy [Esomeprazole, Moxifloxacin, Amoxicillin] — moxifloxacin triple therapy [Esomeprazole, 40 mg bid 7 days (D1-D7)+Moxifloxacin, 400 mg qd 7 days (D1-D7)+Amoxicillin 1 g bid 7 days (D1-D7)].
  Other Names: 7d MEA triple therapy
  Arms: 7 days tailored MEA therapy group
Drug: 7 or 14 days tailored EBMT therapy group (bismuth quadruple therapy) — bismuth quadruple therapy [Esomeprazole, 40 mg bid 7 days (D1-D7)+amoxicillin 1 g bid 7 days (D1-D7)+clarithromycin 500mg bid 7 days (D1-D7)], bismuth quadruple therapy [Esomeprazole, 40 mg bid 7 days (D1-D7)+Tri potassium dicitrate bismuthate, 300 mg qid 7 days (D1-D7)+Metronidazole, 500 mg tid 7 days (D1-D7)+Tetracycline 500 mg qid 7 days (D1-D7)] If there was no metronidazole resistance, the treatment was 7 days in duration. If metronidazole resistance was evident, treatment duration was 14 days.
  Other Names: 7d or 14d quadruple therapy
  Arms: 7 or 14 days tailored EBMT therapy group

SUMMARY:
To compare the eradication success rate between 10-days sequential therapy and 7-days tailored therapy based on H. pylori culture and antimicrobial susceptibility testing.

DETAILED DESCRIPTION:
As increasing antimicrobial resistance in Korea, the effectiveness of empirical Helicobacter pylori (H. pylori) therapies have been declined. Recently, 10-day sequential therapy was not sufficient to overcome tough situation for H. pylori eradication.

Thus, in this study, the investigators evaluated the efficacy of H. pylori eradication between a 7 days tailored therapy (7 day PPI based triple therapy, bismuth quadruple therapy or moxifloxacin contained triple therapy) for H. pylori infection based on the results of antibiotics resistance by using H. pylori culture and minimal inhibitory concentration (MIC) and the 10 day sequential therapy for the first eradication of H. pylori infection, and the investigators analyzed the prevalence of the antibiotic resistance in the tailored therapy group.

ELIGIBILITY:
Inclusion Criteria:

* The patients who proved H. pylori infection following three methods

  1. positive rapid urease test (CLOtest)
  2. histologic evidence of H. pylori by modified Giemsa staining
  3. positive Urea breath test
* Male and female Korean Adult (Aged ≥ 18 years)

Exclusion Criteria:

* Patients who received eradication therapy for H. pylori infection, previously
* H. pylori eradication failure because of poor compliance
* the administration of antibiotics or the consumption of bismuth salts within 4 weeks or the administration of a proton pump inhibitor (PPI) within 2 weeks
* Advanced gastric cancer or other malignancy
* Abnormal liver function or liver cirrhosis
* Abnormal renal function or chronic kidney disease
* Other severe concurrent diseases
* Previous allergic reactions to the study drugs
* Pregnant or lactating women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-08; Primary Completion 2024-04 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Compare the percentage of participants with successful H. pylori eradication in each groups | 6 weeks after completion of eradication
  The efficacy of H. pylori eradication between a 7 days tailored therapy for H. pylori infection based on the results of antimicrobial resistance by using H. pylori culture and minimal inhibitory concentration (MIC) and the 10 days therapy as first eradication regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Nayoung Kim, M.D., Ph. D, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea